CLINICAL TRIAL: NCT06385535
Title: Clinical Characteristics and Temporal Properties of Individual Tics in Persistent Tic Disorder
Acronym: PTD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Kirsten Bootes, Clinical Psychology Doctoral Candidate, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB_00171031
Record Dates: First submitted 2024-01-30; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Tics; Tic Disorders; Vocal Tic; Motor Tic; Tourette Syndrome; Tourette Syndrome in Children; Tourette Syndrome in Adolescence; Tics/Tremor
Keywords: Tics; Tic Disorders; Vocal Tic; Motor Tic; Tourette Syndrome; Tourette Syndrome in Children; Tourette Syndrome in Adolescence; Tics/Tremor
MeSH Terms: conditions — Tics; Tic Disorders; Tourette Syndrome | interventions — Therapeutics; Behavior Therapy

STUDY DESIGN:
Intervention Model Description: Clinical trial with a single arm (i.e., participants are not assigned to groups).
Masking Description: The Principal Investigator and Outcomes Assessors will be blinded to the fractal properties of participants' tics until all study procedures have been completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Habit Reversal Training (HRT) (Experimental): All participants receive 4 sessions of HRT (Habit Reversal Training) to treat their tics.
  Interventions: Behavioral: Habit Reversal Training (HRT)

INTERVENTIONS:
Behavioral: Habit Reversal Training (HRT) — Habit Reversal Training (HRT) is a multicomponent treatment package developed to treat a repetitive behaviors. HRT includes (1) increasing awareness of discrete occurrences of tics and associated premonitory urges (PMUs; i.e., awareness training), (2) teaching the patient to suppress tics by engaging in behaviors that are physically incompatible with target tics (i.e., competing response [CR] training), and (3) prompting and reinforcing between-session patient engagement with therapeutic techniques and homework (i.e., providing social support).
  Other Names: Therapy; Behavior Therapy; Comprehensive Behavioral Intervention for Tics; CBIT; Habit Reversal Therapy; HRT; Tic Therapy

SUMMARY:
The goal of this clinical study is to learn more about the timing of tics (sudden, fast movements and sounds that people do and make without meaning to) in people who have multiple tics that have been going on for more than one year. The main questions it aims to answer are:

1. See whether a tic's timing is related to other characteristics of the tic, like how long it has been happening and how well the person can control/stop that tic
2. See whether the timing of a tic can tell us how well the person can control/stop that tic
3. See whether tic treatment changes the timing of tics, and if the timing of a tic has anything to do with how well treatment will work to stop it

Participants will meet with a study researcher to learn more about the study, ask questions, and decide whether or not they would like to be involved. If they decide to do the study, they will meet with the researcher 6 times:

1. During the first visit, the study researcher will ask questions about the participant's life, tics, and other psychological symptoms. The researcher will watch the participant's tics for 10 minutes. The participant will do a computer task where they follow instructions to tic or not tic.
2. During the second visit, the study researcher will treat one of the participant's tics.
3. During the third visit, the study researcher will treat another one of the participant's tics.
4. During the fourth visit, the study researcher will treat another one of the participant's tics.
5. During the fifth visit, the study researcher will treat another one of the participant's tics.
6. During the sixth visit, the study researcher will ask questions about the participant's tics and other psychological symptoms. The participant will do a computer task where they follow instructions to tic or not tic.

DETAILED DESCRIPTION:
Interested participants will attend an initial phone call or virtual meeting to explain the study, answer any study-related questions, and screen for eligibility.

The consent and assent process will take place online via secure videoconference. Parents will be instructed ahead of time to be in a secure location with their child. Study personnel will explain the study, review the parental permission/consent and assent forms, and answer study-related questions. Participants will be asked to consider and discuss study participation with the study personnel out of the virtual room to encourage the participants to discuss his/her/their willingness to participate and any concerns that they may have. Children will also be asked to provide verbal assent/willingness to participate during this process. If the child is unsure at that time, he/she/they will be encouraged to ask questions and for the parents to reach out again in the future if the child would like to provide verbal assent or decline to participate.

All study visits will take place online via secure videoconference and be video recorded and later coded for reliability and procedural fidelity. Participation will involve six visits that comprise three phases: 1) a pre-treatment (baseline) assessment; 2) four sessions of standard Habit Reversal Training (HRT) for tics, and 3) a post-treatment assessment. At the beginning of the HRT visits, participants will also undergo a direct observation of their tics. At the beginning of the baseline and post-assessment visits, participants will also undergo a standard reinforced tic suppression task (RTST) consisting of three repeated alterations (ABABAB) of a free-to-tic (FTT; A condition) and a differential reinforcement for tic suppression condition (DRO; B condition). Participants who withdraw from the study before their post-treatment assessment will be asked to attend a final study visit to document their reason for withdrawal and complete the debriefing process, however, this visit will be voluntary. All measures aside from the demographics form and between-session activities form are standardized.

Study Visit #1 (Phase 1: Pre-Treatment [Baseline] Assessment)

Following the informed consent/assent process, families will complete a clinical interview with trained study personnel. The clinical interview will confirm that the participant meets the criteria for the study and collect information for subsequent study procedures. Then, the child participant will engage in the RTST. Overall, the first study visit will take approximately 2 hours to complete.

Clinical Interview and Assessment: The clinical interview will include general questions regarding the child's tic symptoms and other psychological/behavioral symptoms/disorders, overall functioning, and family medical history. The diagnostic assessment will consist of the Yale Global Tic Severity Scale (YGTSS) to determine overall tic severity and obtain a list of operationally-defined tics; the Parent Tic Questionnaire (PTQ) to determine individual tic severity; and the Individualized Premonitory Urge for Tics Scale (I-PUTS) to characterize general and individual premonitory urge severity of tics, respectively. The clinical interview will also include a 10-minute tic observation period.

History and Demographics Form: Parents will complete a demographic form collecting data about age, gender, race/ethnicity, occupational/educational history, psychiatric and medical status/history, treatment history and medication status, and other relevant psychosocial factors.

Tic Observation: The child will be directly observed for 10 minutes with the study personnel off-camera to ensure that they meet the criteria for enrollment (i.e., display at least four different tics per minute, on average).

Reinforced Tic Suppression Task (RTST)

The RTST will be comprised of repeated sessions of two experimental conditions: FTT (Condition A) and DRO (Condition B). Each condition will be repeated three times for a total of six sessions (ABABAB). Each session will last 5 minutes, and the order of sessions will be identical across all participants and administrations. During each session, participants will be seated facing their computer's video camera. The child will be provided with specific instructions for the condition and an investigator will monitor the child's performance covertly (via video) to ensure procedural adherence during the session. A manipulation check will be conducted immediately after each session, during which the participant will be asked to repeat the instructions that they were given for the recently completed session and rate how hard they tried to suppress their tics and how well they thought they suppressed their tics. For the DRO conditions, participants will also be asked how they earned tokens.

FTT condition 1A. The purpose of this condition is to establish tic rate in the absence of reinforcement and will serve as a comparison for the DRO condition described below. In the FTT condition, participants will be told that they should feel free to tic as little or as much as they need to, but to avoid suppressing their tics. No reinforcement will be delivered during this condition.

DRO condition 1B. The purpose of this condition is to examine the effects of differential reinforcement on tic frequency. Prior to the start of the condition, participants will be instructed to suppress their tics and will be informed that they will earn a token for every 10-second interval (i.e., trial) in which they do not display any tics. The experimenter will monitor tics and deliver reinforcers by displaying a digital image of a token on the child's screen according to a resetting DRO 10-s schedule, wherein a token will be delivered immediately after each trial during which no tics are observed. If one or more tics are observed during a trial, reinforcement will be withheld, and the count-down timer will be reset.

FTT conditions 2A and 3A. The third and fifth sessions will involve repetitions of the FTT 1A condition described above.

DRO conditions 2B and 3B. The fourth and sixth sessions will involve repetitions of the DRO 1B condition described above.

Study Visits #2-5 (Phase 2: Habit Reversal Training [HRT])

Participants will engage in four HRT sessions delivered across five weeks via secure videoconference. Each session of HRT will be focused on a single, target tic. The target tic for each HRT session will be predetermined following the baseline assessment and before the first session of HRT. The target tics will be randomly chosen from a subset of a list of operationally defined tics that are hierarchically arranged by frequency based on the results obtained from the YGTSS and PTQ administered at the baseline assessment. If, during the study, participants report newly onset tics, they will be documented but will not be targeted in treatment.

To assess between-session differences across participants, HRT sessions 2-4 will begin with participants answering questions about between-session HRT practice. Next, a 10-minute direct observation of tics will be conducted to determine the resting tic rate. The child will be instructed to feel free to tic as little or as much as they need but to avoid suppressing their tics. Participants will then engage in brief HRT for a single, target tic consistent with manualized procedures. HRT will begin with awareness training, including developing a detailed description of the target tic and practicing "catching" the target tic before it occurs. Participants will engage in this exercise for 10 minutes or until they can successfully catch their target tic at least 80% of the time that it occurs within a five-minute period, whichever occurs first. The participant will then engage in competing response (CR) training, including identifying a behavior that can be observed and is incompatible with the target tic. Participants will be instructed to engage in that behavior when they feel the urge associated with their target tic for one minute, or until the urge subsides, whichever is longer. Participants will be verbally prompted by the therapist to engage in the CR whenever the target tic is observed. Participants will practice using the selected CR to suppress their target tic for 10 minutes or until they can use it effectively at least 80% of the time over a five-minute period, whichever occurs first. The participant will be instructed to engage in 15 minutes of CR practice for their target tic(s) each day before the next treatment session. Parents of participants will be instructed to partake in the daily CR practice session with their child by prompting and verbally reinforcing the use of the CR. Overall, the approximate duration of treatment sessions will be 45 to 60 minutes.

Study Visit #6 (Phase 3: Post-Treatment Assessment)

The post-treatment assessment will occur within one week of the last HRT session. To assess between-session differences across participants, the post-treatment assessment will begin with participants answering a series of questions regarding between-session practice and adverse events. Next, participants will engage in the RTST. Participants will then complete a diagnostic assessment with trained study personnel consisting of the YGTSS, PTQ, and I-PUTS. Participation will be considered complete at this point.

ELIGIBILITY:
Inclusion Criteria:

* 8 to 12 years old child who meets the criteria for diagnosis of a persistent tic disorder (e.g., persistent motor/vocal tic disorder or Tourette's disorder; i.e., engages in motor and/or vocal tics that have been present for at least one year)
* The child's tics initially onset before age 10.
* The child currently engages in at least four different motor and/or vocal tics per minute, on average, during a 10-minute observation period.
* The child has a minimum Total Tic Severity Score of 20 on the Yale Global Tic Severity Scale (10 for motor or vocal tics only)
* If the child is on tic-suppressing or psychotropic medication, the dose has been stable for at least 6 weeks with no changes or planned changes in medication status during the study period.
* Parent and child read and speak fluent English.
* The parent is 18+ years of age.
* Access to a private computer with high-speed internet access and private setting.

Exclusion Criteria:

* If, based on the assessment of the study investigators, the child has any serious psychiatric or neurological condition that would interfere with study participation (e.g., unmanaged attention-deficit hyperactivity disorder)
* The child has a self- or parent-reported history of, or is reasonably suspected to have or meet criteria for, functional neurological symptom disorder.
* The child has received more than two sessions of behavioral treatment for tics for which tic suppression was a primary component.
* The child has a Total Tic Severity Score of 40+ on the Yale Global Tic Severity Scale (20+ for motor/vocal tics only).

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Estimates of baseline individual and total tic fractality within free-to-tic (FTT) and differential reinforcement of other behavior (DRO) environmental contingencies | Pre-intervention (baseline)
  Estimates of individual and total tic fractality at baseline will be obtained using tic time series data (i.e., temporal sequences of the presence or absence of tics) during the three free-to-tic (FTT) and three differential reinforcement of other behavior (DRO) conditions of the reinforced tic suppression task (RTST) administered at baseline (pre-intervention). The degree to which individual and total tic time series' follow the frequency spectrum of pink noise (R^2i) will be calculated and conditionally aggregated to provide average estimated fractal exponents.
Voluntary tic suppression success at baseline | Pre-intervention (baseline)
  Voluntary individual and total tic suppression success will be measured by the average proportion of change of individual and total tic frequency from the three free-to-tic (FTT) and three differential reinforcement of other behavior (DRO) conditions of the reinforced tic suppression task (RTST) administered at baseline. Larger differences between the average number of tics observed during FTT and DRO conditions will indicate greater voluntary suppression success.
Total tic severity at baseline as measured by the Yale Global Tic Severity Scale (YGTSS) | Pre-intervention (baseline)
  The Yale Global Tic Severity Scale (YGTSS) will be used to measure total tic severity at baseline across five dimensions: number, frequency, intensity, complexity, and interference. Scores range from 0-5 (low-high) on each dimension and are totaled to indicate overall severity during the past week. Scores are summed to provide a Total Tic Severity Score ranging from 0-50 (none-severe).
Total and individual tic severity at baseline as measured by the Parent Tic Questionnaire (PTQ) | Pre-intervention (baseline)
  The Parent Tic Questionnaire (PTQ) will be used to characterize individual and total tic severity at baseline. The PTQ assesses for the presence of common motor and vocal tics over the past week. Frequency and intensity scores ranging from 1-4 (low, high) are obtained for each endorsed tic, which can be summed to yield an individual tic severity score ranging from 0-8 (low, high).
Changes in voluntary individual and total tic suppression success pre- and post-intervention | Pre-intervention (baseline), up to 1 week post intervention
  Voluntary individual and total tic suppression success will be measured by the average proportion of change of individual and total tic frequency from the three free-to-tic (FTT) and three differential reinforcement of other behavior (DRO) conditions of the reinforced tic suppression tasks (RTSTs) administered at baseline and post-treatment. Larger differences between the average number of tics observed during FTT and DRO conditions at individual time points will indicate greater voluntary suppression success. Larger differences between estimates of suppression success before and after HRT will indicate greater changes in suppression abilities following treatment.
Changes in individual and total tic fractality within free-to-tic (FTT) and differential reinforcement of other behavior (DRO) environmental contingencies pre- and post-intervention | Pre-intervention (baseline), up to 1 week post intervention
  Estimates of individual and total tic fractality at baseline and post-intervention will be obtained using tic time series data (i.e., temporal sequences of the presence or absence of tics) during the three free-to-tic (FTT) and three differential reinforcement of other behavior (DRO) conditions of the reinforced tic suppression task (RTST) administered at baseline (pre-intervention) and post-intervention, respectively. The degree to which individual and total tic time series' follow the frequency spectrum of pink noise (R^2i) will be calculated and conditionally aggregated to provide average estimated fractal exponents at individual time points. Larger differences between fractal exponents before and after HRT will indicate greater changes in tic fractality following treatment.
Changes in individual and total tic severity pre- and post-intervention as measured by the Yale Global Tic Severity Scale (YGTSS) and Parent Tic Questionnaire (PTQ) | Pre-intervention (baseline), up to 1 week post intervention
  The Yale Global Tic Severity Scale (YGTSS) measures total tic severity across five dimensions: number, frequency, intensity, complexity, and interference. Scores range from 0-5 (low-high) on each dimension and are totaled to indicate overall severity during the past week. Scores are summed to provide a Total Tic Severity Score ranging from 0-50 (none-severe). The Parent Tic Questionnaire (PTQ) measures individual and total tic severity by assessing for the presence of common motor and vocal tics over the past week. Frequency and intensity scores ranging from 1-4 (low, high) are obtained for each endorsed tic, which can be summed to yield an individual tic severity score ranging from 0-8 (low, high). The YGTSS and PTQ will be used to measure total and individual and total tic severity, respectively, at baseline and post-intervention. Larger differences between YGTSS and PTQ scores before and after HRT will indicate greater changes in tic severity following treatment.

SECONDARY OUTCOMES:
Individual and total premonitory urge severity at baseline as measured by the Individualized Premonitory Urge for Tics Scale (I-PUTS) | Pre-intervention (baseline)
  The Individualized Premonitory Urge for Tics Scale (I-PUTS) is a clinician-administered measure of the frequency and intensity of premonitory urges associated with individual tics that will be used to characterize individual and total premonitory urge severity at baseline. Scores ranging from 1-4 (almost never-frequent; minimal-strong) on each dimension are totaled to produce a Total Urge Intensity and Frequency score.
Individual and total premonitory urge severity post-intervention as measured by the Individualized Premonitory Urge for Tics Scale (I-PUTS) | Up to 1 week post intervention
  The Individualized Premonitory Urge for Tics Scale (I-PUTS) is a clinician-administered measure of the frequency and intensity of premonitory urges associated with individual tics that will be used to characterize individual and total premonitory urge severity post-intervention. Scores ranging from 1-4 (almost never-frequent; minimal-strong) on each dimension are totaled to produce a Total Urge Intensity and Frequency score.
Changes in individual and total premonitory urge severity pre- and post-intervention as measured by the Individualized Premonitory Urge for Tics Scale (I-PUTS) | Pre-intervention (baseline), up to 1 week post intervention
  The Individualized Premonitory Urge for Tics Scale (I-PUTS) is a clinician-administered measure of the frequency and intensity of premonitory urges associated with individual tics that will be used to characterize individual and total premonitory urge severity at baseline and post-intervention. Scores ranging from 1-4 (almost never-frequent; minimal-strong) on each dimension are totaled to produce a Total Urge Intensity and Frequency score. Larger differences between total and individual tic I-PUTS scores before and after HRT will indicate greater changes in premonitory urge severity following treatment.
Total tic severity post-intervention as measured by the Yale Global Tic Severity Scale (YGTSS) | Up to 1 week post intervention
  The Yale Global Tic Severity Scale (YGTSS) will be used to measure total tic severity post-intervention across five dimensions: number, frequency, intensity, complexity, and interference. Scores range from 0-5 (low-high) on each dimension and are totaled to indicate overall severity during the past week. Scores are summed to provide a Total Tic Severity Score ranging from 0-50 (none-severe).
Individual and total tic severity post-intervention as measured by the Parent Tic Questionnaire (PTQ) | Up to 1 week post intervention
  The Parent Tic Questionnaire (PTQ) will be used to characterize individual and total tic severity at baseline. The PTQ assesses for the presence of common motor and vocal tics over the past week. Frequency and intensity scores ranging from 1-4 (low, high) are obtained for each endorsed tic, which can be summed to yield an individual tic severity score ranging from 0-8 (low, high).
Voluntary tic suppression success post-intervention | Up to 1 week post intervention
  Voluntary individual and total tic suppression success will be measured by the average proportion of change of individual and total tic frequency from the three free-to-tic (FTT) and three differential reinforcement of other behavior (DRO) conditions of the reinforced tic suppression task (RTST) administered post-intervention. Larger differences between the average number of tics observed during FTT and DRO conditions will indicate greater voluntary suppression success.
Estimates of individual and total tic fractality within free-to-tic (FTT) and differential reinforcement of other behavior (DRO) environmental contingencies post-intervention | Up to 1 week post intervention
  Estimates of individual and total tic fractality post-intervention will be obtained using tic time series data (i.e., temporal sequences of the presence or absence of tics) during the three free-to-tic (FTT) and three differential reinforcement of other behavior (DRO) conditions of the reinforced tic suppression task (RTST) administered post-intervention. The degree to which individual and total tic time series' follow the frequency spectrum of pink noise (R^2i) will be calculated and conditionally aggregated to provide average estimated fractal exponents.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Himle, PhD, Study Chair — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in any publication(s) may be provided to qualified researchers. All data shared will be coded with no identifying information included. Approval of the request by the study primary investigator and execution of all applicable data sharing agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after publication.
Access Criteria: Qualified researchers are those considered to have academic interests in tic disorders and related conditions, expertise in the scoring and interpretation of the outcome measures administered, and a reasonable and scientifically-sound justification for obtaining participant data.

REFERENCES:
- [Background] Woods DW, Himle MB. Creating tic suppression: comparing the effects of verbal instruction to differential reinforcement. J Appl Behav Anal. 2004 Fall;37(3):417-20. doi: 10.1901/jaba.2004.37-417. PMID 15529900
- [Background] Leckman JF, Riddle MA, Hardin MT, Ort SI, Swartz KL, Stevenson J, Cohen DJ. The Yale Global Tic Severity Scale: initial testing of a clinician-rated scale of tic severity. J Am Acad Child Adolesc Psychiatry. 1989 Jul;28(4):566-73. doi: 10.1097/00004583-198907000-00015. PMID 2768151
- [Background] McGuire JF, McBride N, Piacentini J, Johnco C, Lewin AB, Murphy TK, Storch EA. The premonitory urge revisited: An individualized premonitory urge for tics scale. J Psychiatr Res. 2016 Dec;83:176-183. doi: 10.1016/j.jpsychires.2016.09.007. Epub 2016 Sep 9. PMID 27643476
- [Background] Storch EA, Murphy TK, Geffken GR, Sajid M, Allen P, Roberti JW, Goodman WK. Reliability and validity of the Yale Global Tic Severity Scale. Psychol Assess. 2005 Dec;17(4):486-91. doi: 10.1037/1040-3590.17.4.486. PMID 16393016
- [Background] Azrin NH, Nunn RG. Habit-reversal: a method of eliminating nervous habits and tics. Behav Res Ther. 1973 Nov;11(4):619-28. doi: 10.1016/0005-7967(73)90119-8. No abstract available. PMID 4777653
- [Background] Miltenberger RG, Fuqua RW. A comparison of contingent vs non-contingent competing response practice in the treatment of nervous habits. J Behav Ther Exp Psychiatry. 1985 Sep;16(3):195-200. doi: 10.1016/0005-7916(85)90063-1. PMID 4066967
- [Background] Chang S, Himle MB, Tucker BTP, Woods DW, Piacentini J. Initial psychometric properties of a brief parent-reported instrument for assessing tic severity in children with chronic tic disorders. Child & Family Behavior Therapy. 2009;31:181-191.

DOCUMENTS (1):
  • Informed Consent Form (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/35/NCT06385535/ICF_000.pdf